CLINICAL TRIAL: NCT04603378
Title: A Randomized, Double-blind, Placebo-controlled Study to Evaluate the Effect of Novel Glycans on Nitrogen Metabolism of the Gut in Healthy Subjects Using a Stable Isotope
Brief Title: A Clinical Study to Assess the Effect of Novel Glycans on Nitrogen Metabolism of the Gut in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kaleido Biosciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: K010-117
Record Dates: First submitted 2020-10-21; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Healthy
Keywords: microbiome; nitrogen metabolism; Kaleido; Kaleido Biosciences; KB195; Oligosaccharide; Glycan; Microbiome metabolic therapy; MMT
MeSH Terms: interventions — polydextrose; pullulan; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- KB195 (Other)
  Interventions: Other: KB195
- Polydextrose (Other)
  Interventions: Other: Polydextrose
- Pullulan (Other)
  Interventions: Other: Pullulan
- Maltodextrin (Other)
  Interventions: Other: Maltodextrin

INTERVENTIONS:
Other: KB195 — KB195 is a novel glycan
  Arms: KB195
Other: Polydextrose — Polydextrose is an oligosaccharide
  Arms: Polydextrose
Other: Pullulan — Pullulan is an oligosaccharide
  Arms: Pullulan
Other: Maltodextrin — Maltodextrin is a digestible carbohydrate
  Arms: Maltodextrin

SUMMARY:
This exploratory, randomized, double-blind, placebo-controlled study aims to explore the effect of novel glycans on nitrogen metabolism in the gut in healthy subjects using a stable isotope.

ELIGIBILITY:
To be eligible for inclusion, the patient must fulfill all of the following criteria at screening:

* Willing to provide multiple stool samples
* Be male or female, ≥18 and <50 years of age
* Have a body mass index ≥18 and <50 kg/m2
* No current renal, hepatic or metabolic disease, significant dyslipidemia, or infection
* Willing to adhere to dietary requirements as stated in the protocol
* Willing to continue usual exercise routine
* Willing to continue taking any current supplements and vitamins (with the exception of prebiotic or probiotic supplements) that the subject is currently taking, for the duration of the study

Patients will be excluded from the study if they meet any of the following criteria at screening :

* Currently taking probiotic or prebiotic dietary supplements, or have taken them in the past 28 days (prior to Screening Visit), or unwilling to avoid prebiotic or probiotic dietary supplements for the duration of the study
* Currently taking, or have taken during the last seven days prior to enrollment, drugs or other compounds that modulate GI motility
* Currently taking bismuth, or have taken bismuth within seven days prior to enrollment
* Recent history (within six weeks of Screening Visit) of the following condition requiring medical attention or treatment, including over-the-counter medications: constipation, diarrhea, and/or acute GI illness.
* Systemic antibiotics taken within the previous three months (prior to Screening Visit).
* History of or active inflammatory bowel disease
* History of or active irritable bowel syndrome
* History of or active autoimmune disease.
* History of or active GI malignancy.
* Established pre-diabetic status (eg, multiple fasting blood glucose measurements 100 to 125 mg/dL inclusive, or history of failed glucose tolerance tests) and as assessed by HbA1c test.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 47 (Actual)
Dates: Start 2017-09-18 (Actual); Primary Completion 2017-11-28 (Actual); Study Completion 2017-11-28 (Actual)

PRIMARY OUTCOMES:
Number of patients experiencing any treatment-emergent adverse events (TEAEs) | Day -8 to Day 29

CONTACTS AND LOCATIONS:
Overall Officials: Mark Wingertzahn, PhD, Study Director — Kaleido Biosciences
Locations (1):
- PPD Phase I Clinic, Austin, Texas, United States